CLINICAL TRIAL: NCT04533386
Title: A Multicomponent Intervention to Increase HIV Risk Perceptions and PrEP Initiation Among Black Men Who Have Sex With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Derek Dangerfield II, PI, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00241244
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: HIV Risk Perception; PrEP

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BSMM (Experimental): Intervention arm will include motivational interview-consistent discussion with a peer change agent and use of a mobile application to record and review sexual risk behaviors with participants.
  Interventions: Behavioral: Multi-component intervention strategy

INTERVENTIONS:
Behavioral: Multi-component intervention strategy — Multi-component intervention strategy using a peer change agent and mobile application to record and review sexual risk behaviors

SUMMARY:
Tragically, HIV infections among Black sexual minority men (BSMM) in the U.S. persist. Despite the availability of pre-exposure prophylaxis (PrEP) for HIV prevention, effective uptake among BSMM remains low. It is imperative to support PrEP initiation among this group. The proposed multi-component interventional study is designed to increase HIV risk perceptions and subsequent PrEP initiation through the use of our team's existing mobile application called PrEPme and a peer change agent (PCA) to record and review sexual risk behaviors and subsequent PrEP interest. Few have studied whether reviewing sexual diaries with a PCA increases HIV risk perceptions and PrEP initiation among BSMM. This strategy will allow BSMM who are not using PrEP to record their sexual behaviors using a PrEPme-based diary, review their sexual histories with a PCA, and assess PrEP interest. The PCA will be trained in motivational interviewing techniques to facilitate discussions. The PCA will provide HIV prevention education, sexual risk evaluation, and PrEP navigation. BSMM who become interested in initiating PrEP will be referred to our team's ongoing PrEP tele-medicine study (PI: Jason Farley, co-investigator) or other PrEP care services in the greater Baltimore area. The proposed intervention targets a high priority population in HIV prevention and mitigates structural barriers to PrEP uptake such as perceived judgement, stigma, and discrimination from clinical providers.

DETAILED DESCRIPTION:
The proposed multicomponent intervention will use our team's existing mobile smartphone app called PrEPme along with a peer change agent (PCA) to record and review sexual risk behaviors among 80 HIV-negative BSMM. PrEPme is an existing HIPAA compliant mobile app that is currently available in the mobile application "store" and offers PrEP navigation services in Baltimore and throughout the State of Maryland. Currently, the app contains a diary that allows users to record and review their sexual risk behaviors using a weekly "timeline" including number and gender of partners along with substance use. At the end of each week, the dashboard provides a weekly review of sexual history for four weeks until the history is displayed as a monthly overview. The app also allows users to chat with our case management team to learn more about PrEP, obtain adequate insurance coverage, and get help scheduling appointments at any time. The proposed intervention leverages the current features of the app as part of the multi-component strategy. In the intervention, pre-post assessments will include demographic information, sexual behavior, substance use, mental health (e.g., depression, gay community affiliation), and PrEP use history. HIV risk perception will be measured using an 8-item scale. The PCA will be trained to review sexual histories, highlight HIV and sexually transmitted infection risks, provide HIV prevalence information, deliver PrEP information, and encourage PrEP uptake. This intervention phase will use a single-group pretest post-test design to explore feasibility and findings will be used as the foundation for an efficacy trial among a larger sample of BSMM in different locales.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Identify as cis-gender man
* Self-reporting being HIV-negative or status unknown
* Identify as Black or African American
* Report anal intercourse with ≥ 1 male partner in the past 12 months
* Has mobile smartphone
* Not currently taking Truvada or Descovy as pre-exposure prophylaxis (PrEP)

Exclusion Criteria:

* ≤18 years of age
* Identify as woman or transgender
* Self-reporting being HIV-positive
* Identify as race/ethnicity other than Black or African American
* Report no anal intercourse with male partner in the past 12 months
* Report not having a mobile smartphone
* Currently taking Truvada or Descovy as pre-exposure prophylaxis (PrEP)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cis-gender men
Enrollment: 69 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
HIV risk perception as assessed by the Perceived Risk of HIV Scale | 1 month
  The Perceived Risk of HIV Scale is an 8-item scale with each item being scored from 1-5 (e.g., "Extremely likely" to "Extremely Unlikely," "Rarely" to "All of the time," etc.). Overall score ranges from 10 to 40 where higher scores signify increased perception of risk.

SECONDARY OUTCOMES:
Proportion of participants who express interest in PrEP initiation | 1 month
  The proportion of participants who express interest in initiating PrEP at month 1 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Dangerfield II, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young LE, Schumm P, Alon L, Bouris A, Ferreira M, Hill B, Khanna AS, Valente TW, Schneider JA. PrEP Chicago: A randomized controlled peer change agent intervention to promote the adoption of pre-exposure prophylaxis for HIV prevention among young Black men who have sex with men. Clin Trials. 2018 Feb;15(1):44-52. doi: 10.1177/1740774517730012. Epub 2017 Sep 1. PMID 28862483
- [Background] Napper LE, Fisher DG, Reynolds GL. Development of the perceived risk of HIV scale. AIDS Behav. 2012 May;16(4):1075-83. doi: 10.1007/s10461-011-0003-2. PMID 21785873
- [Background] Dangerfield Ii DT, Harawa NT, McWells C, Hilliard C, Bluthenthal RN. Exploring the preferences of a culturally congruent, peer-based HIV prevention intervention for black men who have sex with men. Sex Health. 2018 Nov;15(5):424-430. doi: 10.1071/SH18057. PMID 30185352
- [Derived] Dangerfield Ii DT, Anderson JN, Wylie C, Bluthenthal R, Beyrer C, Farley JE. A Multicomponent Intervention (POSSIBLE) to Improve Perceived Risk for HIV Among Black Sexual Minority Men: Feasibility and Preliminary Effectiveness Pilot Study. JMIR Hum Factors. 2024 Jun 11;11:e54739. doi: 10.2196/54739. PMID 38861707